CLINICAL TRIAL: NCT05373264
Title: HYDROchlorothiazide to PROTECT Polycystic Kidney Disease Patients and Improve Their Quality of Life
Acronym: HYDRO-PROTECT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Ron Gansevoort, Prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100714; 2021-005612-61 (EudraCT Number)
Record Dates: First submitted 2022-04-28; First posted 2022-05-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: ADPKD
Keywords: ADPKD; Tolvaptan; Hydrochlorothiazide; Quality of Life; Side effects; Polyuria
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polyuria | interventions — Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: An investigator driven, multicenter, placebo-controlled, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrochlorothiazide (Active Comparator): Oral hydrochlorothiazide 25mg, once daily, for a total of 156 weeks
  Interventions: Drug: Hydrochlorothiazide 25 mg
- Placebo (Placebo Comparator): Matching oral placebo, once daily, for a total of 156 weeks. The placebo is inert.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrochlorothiazide 25 mg — An oral capsule containing 25mg of hydrochlorothiazide
  Arms: Hydrochlorothiazide
Drug: Placebo — A matching oral capsule containing placebo
  Arms: Placebo

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is characterized by progressive formation of renal cysts which ultimately lead to a loss of renal function.

Tolvaptan (a V2R antagonist) is currently the only effective treatment for preserving renal function in ADPKD. However, side-effects such as polyuria limit its tolerability and thereby the therapeutic potential. This study will test whether co-administration with hydochlorothiazide can improve V2RA efficacy (slowing kidney function decline) and tolerability (quality of life) in ADPKD. Approximately 300 patients will be enrolled.

DETAILED DESCRIPTION:
Aims: The main objectives of the current study are to prospectively test whether HCT co-treatment can improve V2RA efficacy (slowing kidney function decline) and tolerability (quality of life) in PKD.

Study design: Investigator driven randomized placebo-controlled multicenter trial

Study population: 300 ADPKD patients of ≥18 years, with an eGFR of > 25 mL/min/1.73m2, on stable treatment with the highest tolerated dose of V2RA

Intervention: Oral HCT 25 mg once daily or matching placebo for a total of 156 weeks. The randomization ratio will be 1:1.

Study visit schedule: study measurements will be performed during 12-weekly visits (which is routine care for V2RA treated patients), except for one additional study visit (or telephone call) 2 weeks after the start of treatment

Primary study outcome: Slope of kidney function decline (measured by eGFR)

ELIGIBILITY:
Inclusion Criteria:

* ADPKD diagnosis (modified Ravine criteria)
* ≥18 years old
* eGFR > 25 mL/min/1.73m2
* On stable treatment with the highest tolerated dose of V2RA for a minimum of 3 months

Exclusion Criteria:

* Known intolerance to hydrochlorothiazide
* Use of any diuretic
* Orthostatic hypotension complaints or blood pressure <105/65mmHg during screening visit
* Uncontrolled hypertension (blood pressure >160/100mmHg)
* Hypokalemia (<3.5 mmol/L)
* History of active gout on maintenance preventive treatment for gout (allopurinol, desuric and/or colchicine), defined as ≥2 episodes during the last year
* History of skin cancer (basal cell, squamous cell and melanoma)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Changes in kidney function decline | 156 weeks
  The primary outcome is the change in kidney function decline (assessed as eGFR slope, in ml/min/1.73 m2 per year), calculated with linear mixed models, using all available creatinine values from week 12 until end of treatment between the tolvaptan/placebo and tolvaptan/HCT group.

SECONDARY OUTCOMES:
Changes in eGFR from baseline compared to end of study (12 weeks after End of Treatment) | 168 weeks
  A secondary outcome is the change in eGFR from baseline compared to end of study (12 weeks after end of treatment)
Incidence of 30% decrease in eGFR, end stage kidney disease (EKSD) or renal death | 168 weeks
  A secondary outcome is the incidence of a 30% decrease in eGFR, occurrence of end stage kidney disease (EKSD) or renal death during the entire study period (until the end of study (12 weeks after end of treatment)
Changes in 24-hour urine volume | 156 weeks
  A secondary outcome is the change in 24-hour urine volume, measured at baseline, week 12, week 48, week 96 and week 156 (end of treatment)
Quality of life, assessed by the TIPS questionnaire | 156 weeks
  Changes in Quality of Life measured by the Tolvaptan Impact of Polyuria Scale questionnaire (TIPS) at baseline, week 12, week 48, week 96 and week 156 (end of treatment)
Quality of life, assessed by the ADPKD-UIS questionnaire | 156 weeks
  Changes in Quality of Life measured by the ADPKD-Urinary Impact Scale questionnaire (ADPKD-UIS) at baseline, week 12, week 48, week 96 and week 156 (end of treatment)
Quality of life, assessed by the SF-12 questionnaire | 156 weeks
  Changes in Quality of Life measured by the Short Form 12 questionnaire (SF-12) at baseline, week 12, week 48, week 96 and week 156 (end of treatment)
Quality of life, assessed by the EQ-5D questionnaire | 156 weeks
  Changes in Quality of Life measured by the EuroQol-5 Dimension questionnaire (EQ-5D) at baseline, week 12, week 48, week 96 and week 156 (end of treatment)
Change in V2RA dose | 168 weeks
  V2RA dose during each study visit and compared at the end of study visit (12 weeks after end of treatment) between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group
Change in V2RA discontinuation rate | 168 weeks
  The V2RA discontinuation rate will be compared at the end of study visit (12 weeks after end of treatment) between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group
Changes in serum sodium concentration | 168 weeks
  Changes in serum sodium concentration between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group, measured from baseline until the end of study (12 weeks after end of treatment)
Changes in serum potassium concentration | 168 weeks
  Changes in serum potassium concentration between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group, measured from baseline until the end of study (12 weeks after end of treatment)
Changes in plasma serum calcium concentration | 168 weeks
  Changes in plasma serum calcium concentration between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group, measured from baseline until the end of study (12 weeks after end of treatment)
Changes in serum phosphate concentration | 168 weeks
  Changes in serum phosphate concentration between tolvaptan/placebo and tolvaptan/hydrochlorothiazide group, measured from baseline until the end of study (12 weeks after end of treatment)
Incidence of (serious) adverse events | 168 weeks
  Incidence of (serious) adverse events from baseline until the end of study (12 weeks after end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. R.T. Gansevoort, Principal Investigator — University Medical Center Groningen
Locations (13):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Leuven, Leuven
- France (2):
  - Hospital La Cavale Blanche, Brest
  - Necker-Enfants Malades Hospital, Paris
- Germany (3):
  - Charité University Hospital, Berlin
  - University Hospital Cologne, Cologne
  - Med. Klinik und Poliklinik III, Universitätsklinikum Dresden., Dresden
- Netherlands (3):
  - Amsterdam University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus University Medical Center, Rotterdam
- Fundación Puigvert, Barcelona, Spain
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - University of Sheffield Medical School, Sheffield

IPD SHARING:
Plan to Share IPD: No